CLINICAL TRIAL: NCT00001372
Title: Studies of the Pathogenesis and Natural History of Systemic Lupus Erythematosus (SLE)
Brief Title: Study of Systemic Lupus Erythematosus
Status: Recruiting | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940066; 94-AR-0066
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-10-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Longitudinal Study; Natural History; Lupus Nephritis; Lupus; Systemic Lupus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Longitudinal cohort study with affected SLE patients
- 2: Patient relatives
- 3: Unrelated healthy volunteers

SUMMARY:
This protocol will evaluate patients with systemic lupus erythematosus (SLE) and their relatives to learn more about how the disease develops and changes over time. It will also study genetic factors that make a person susceptible to SLE.

Patients 3 years of age and older with known or suspected SLE and their relatives may be eligible for this study. Patients will be evaluated with a medical history and physical examination, blood and urine tests. Other procedures may include:

1. Electrocardiogram
2. 24-hour urine collection
3. Imaging studies, such as chest and joint X-rays, magnetic resonance imaging (MRI) scans, bone scans, and bone densitometry.
4. Questionnaire about the degree of disease activity, and survey of risk factors for disease complications.
5. Apheresis-Collection of plasma (fluid portion of blood) or blood cells for analysis. Whole blood is collected through a needle in an arm vein. The blood circulates through a machine that separates it into its components. The required component (plasma or cells) is removed and the rest of the blood is returned to the body through the same needle or through a second needle in the other arm.
6. Skin biopsy-Removal of a small skin sample for microscopic analysis. An area of skin is numbed with an anesthetic and a small circular portion (about 1/4 inch in diameter) is removed, using a sharp cookie cutter-type instrument.
7. Kidney, bone marrow or other organ biopsy-Removal of a small sample of organ tissue. These biopsies are done only if they can provide information useful in better understanding the disease or making treatment decisions.
8. Genetic studies-Collection of a blood sample for gene testing.

Patients will be followed at least once a year with a brief history and physical examination and routine blood and urine tests. Some patients may be seen more often. Treatment recommendations will be offered to patients' physicians, and patients who are eligible for other research treatment studies will be invited to enroll.

Participating relatives of patients will fill out a brief medical history questionnaire and provide a DNA sample (either a blood sample or tissue swab from the inside of the cheek) for genetic testing.

DETAILED DESCRIPTION:
This research protocol will evaluate subjects with systemic lupus erythematosus (SLE) and their relatives to study the pathogenesis and natural history of the disease and the mechanisms leading to enhanced organ damage. Patients will be evaluated by a history and physical examination and routine laboratory studies will be obtained as needed to assess disease activity or complications of the disease and to monitor for drug-related toxicities. Blood, skin or urine specimens may be requested for research purposes, including genetic studies. In addition, a subset of these patients will undergo several tests to understand the pathogenic changes affecting their blood vessels. Patients who are eligible for other research protocols will be offered the opportunity to participate in these studies by signed informed consent. Any medical care recommended or provided to the patient will be consistent with routine standards of practice and provided in consultation with the patient s referring physician. Blood and urine samples and cardiovascular testing will also be collected or applied to from healthy volunteers for research purposes and to support the identification and validation of new biomarker candidates.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with known or suspected SLE will be evaluated in either the outpatient or inpatient research ward of the Clinical Center as indicated. Patients will not be selected based on age, race or gender. However, due to the nature of the disease, the patient population will not be expected to be evenly distributed, since SLE is predominantly a disease of young females, with increased prevalence in select racial groups, particularly African Americans and Hispanics. First and second-degree relatives of the patient may be recruited in the study for genetic analysis. We will ask for the patient s permission to contact his/her relatives.

* SLE or suspected SLE established by ACR/EULAR or ACR criteria
* Ability to give informed consent
* Adult and minor relatives (first and second degree) of individuals Included in IV-G (only for genetic studies)
* Ability of the patient or minor relative s parents to give informed consent
* Affected individuals age >= 3 years with no upper age limit
* Healthy Volunteers (non-related) age >=18 with no upper age limit
* Healthy Volunteers (first- and second-degree relatives) age >=3 with no upper age limit
* Vascular studies adults only age >=18 with no upper age limit

EXCLUSION CRITERIA:

* Concomitant medical problems which would confound the interpretation of studies gathered by this protocol. Included in this is the presence of HIV in the blood, active malignancies, or other significant medical conditions that may interferes with interpretation of some lupus studies.
* Concomitant medical, surgical or other conditions for which inadequate facilities are available to support their care at NIH
* Inability or unwillingness to comply with follow up requirements (e.g. distance, social, physical limitations)
* Any comorbidity of medical or psychological/psychiatric condition or treatment after reviewing of patients previous or outside medical records, that in the opinion of the Principal Investigator, would exclude the subjects from the research studies (e.g. Patient requiring urgent and/or acute medical care, surgical or other procedures)
* Unwilling to participate in research studies or to provide research samples or data
* Any concomitant medical problems or are taking medications which would confound the interpretation of studies they are considered for

EXCLUSION CRITERIA FOR VASCULAR STUDIES ONLY, FOR SLE AND HEALTHY CONTROLS:

* Subjects with a contraindication to MRI scanning will not receive the optional Cardiovascular MRI. These contraindications include subjects with the following devices:

  * Central nervous system aneurysm clips unless it is labeled safe or conditional for MRI
  * Implanted neural stimulator (e.g.TENS-Unit) unless it is labeled safe or conditional for MRI
  * Implanted cardiac pacemaker or defibrillator unless it is labeled safe or conditional for MRI
  * Cochlear or any type of ear implant unless it is labeled safe or conditional for MRI
  * Ocular foreign body (e.g. metal shavings)
  * Implanted Insulin pump or drug infusion device unless it is labeled safe or conditional for MRI
  * Metal shrapnel or bullet unless cleared by plain x-ray as safe for MRI
* Subjects with renal excretory dysfunction, estimated glomerular filtration rate < 60 mL/min/1.73m^2 using the CKD-EPI equation or equivalent (using the CRIS-calculated eGFR to define the threshold) and a serum creatinine measured within 2 weeks without intercurrent change in medical condition or medications. Subjects meeting this exclusion criterion may still be included in the study but will not be exposed to the cardiac CT angiography, or gadolinium-based contrast agents.
* Pregnant or lactating women will be excluded from vascular studies.
* Any clinical instability precluding subject from getting MRI as determined by the enrolling clinician.
* Healthy controls with known history of coronary artery disease, peripheral vascular disease or atherosclerosis.
* Individuals younger than 18 years old will be excluded given the radiation exposure as well as the lack of proper validation for the proposed vascular function studies.

Ages: 3 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: subjects with systemic lupus erythematosus (SLE) and their relatives
Sampling Method: Non-Probability Sample
Enrollment: 2250 (Estimated)
Dates: Start 1994-02-10 (Actual)

PRIMARY OUTCOMES:
Natural History of SLE | 12/31/2050
  Natural History of SLE

CONTACTS AND LOCATIONS:
Overall Officials: Sarfaraz A Hasni, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We plan to share aggregate data for analysis. Any IPD shared will be deidentified and coded.

REFERENCES:
- [Derived] Lee Y, Wessel AW, Xu J, Reinke JG, Lee E, Kim SM, Hsu AP, Zilberman-Rudenko J, Cao S, Enos C, Brooks SR, Deng Z, Lin B, de Jesus AA, Hupalo DN, Piotto DG, Terreri MT, Dimitriades VR, Dalgard CL, Holland SM, Goldbach-Mansky R, Siegel RM, Hanson EP. Genetically programmed alternative splicing of NEMO mediates an autoinflammatory disease phenotype. J Clin Invest. 2022 Mar 15;132(6):e128808. doi: 10.1172/JCI128808. PMID 35289316
- [Derived] Wu J, Singh K, Lin A, Meadows AM, Wu K, Shing V, Bley M, Hassanzadeh S, Huffstutler RD, Schmidt MS, Blanco LP, Tian R, Brenner C, Pirooznia M, Kaplan MJ, Sack MN. Boosting NAD+ blunts TLR4-induced type I IFN in control and systemic lupus erythematosus monocytes. J Clin Invest. 2022 Mar 1;132(5):e139828. doi: 10.1172/JCI139828. PMID 35025762
- [Derived] Carlucci PM, Purmalek MM, Dey AK, Temesgen-Oyelakin Y, Sakhardande S, Joshi AA, Lerman JB, Fike A, Davis M, Chung JH, Playford MP, Naqi M, Mistry P, Gutierrez-Cruz G, Dell'Orso S, Naz F, Salahuddin T, Natarajan B, Manna Z, Tsai WL, Gupta S, Grayson P, Teague H, Chen MY, Sun HW, Hasni S, Mehta NN, Kaplan MJ. Neutrophil subsets and their gene signature associate with vascular inflammation and coronary atherosclerosis in lupus. JCI Insight. 2018 Apr 19;3(8):e99276. doi: 10.1172/jci.insight.99276. eCollection 2018 Apr 19. PMID 29669944
- [Derived] Pfiffner PB, Oh J, Miller TA, Mandl KD. ClinicalTrials.gov as a data source for semi-automated point-of-care trial eligibility screening. PLoS One. 2014 Oct 21;9(10):e111055. doi: 10.1371/journal.pone.0111055. eCollection 2014. PMID 25334031
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1994-AR-0066.html